CLINICAL TRIAL: NCT01372098
Title: Development and Evaluation of an Intervention for Intimate Partner Violence in the Context of Nurse Home Visits
Brief Title: Nurse-family Partnership (NFP) Curriculum Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Public Health Agency of Canada (PHAC) (Other Government); Annie E. Casey Foundation (Other Government)
Responsible Party: Principal Investigator, Harriet L. MacMillan, Professor of Pediatrics, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MacMillan_NFP_IPVI_RCT
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Domestic Violence
Keywords: Domestic Violence; Spouse Abuse
MeSH Terms: interventions — Neurofilament Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NFP + IPV intervention (Experimental): The protocol for number and timing of visits will be the same for both NFP+IPVI and Standard Care, as follows: weekly for the first four visits, every other week for the remainder of the pregnancy, every week for six weeks in the postpartum and every other week until the infant is 21 months old after which it is once a month for the last three months. We recognize that the intervention might prompt the nurse and mother to alter the regular visit schedule if IPV is present.
  Interventions: Behavioral: NFP + IPV intervention
- NFP (standard care) (No Intervention): The NFP nurses currently receive some training regarding IPV, but it is minimal. Between intake and when the child is 3 months and 12 months old, there is a brief instruction that the nurse assess for IPV. If the client acknowledges current abuse when completing the Abuse Assessment Screen, the nurse should "assist her to evaluate threats to personal safety and make referrals as needed". There is a prompt to be mindful of client safety, and to make referrals as needed.

INTERVENTIONS:
Behavioral: NFP + IPV intervention — The intervention focuses on helping women stay safe in a relationship. Strategies for overcoming barriers to using and accessing community resources and services, and community agency interventions for women exposed to IPV is built into the intervention.
  Arms: NFP + IPV intervention

SUMMARY:
The purpose of this study is to determine whether the Intimate Partner Violence (IPV) intervention in the context of Nurse-Family Partnership (NFP) program improves women's quality of life and reduces violence relative to the NFP alone using a cluster randomized controlled trial. Our hypothesis is that an IPV intervention can be designed that is acceptable to participants in the NFP, feasible to implement, and that this intervention will improve quality of life for women and reduce exposure to violence.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years and older
* NFP program participants (woman with first live birth and living in poverty)
* English speaker

Exclusion Criteria:

- Woman who cannot communicate in English

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in WHO Quality of Life-BREF at 6, 12, 18, and 24 months | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum

SECONDARY OUTCOMES:
The Composite Abuse Scale (CAS) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Validated 30-item research instrument that assesses exposure to physical, sexual and emotional abuse, harassment and combined severe abuse.
The Domestic Violence Survivor Assessment (DVSA) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Based on Prochaska's Transtheoretical Model of Behaviour Change (also known as "stages of change") and was developed by Dienemann and colleagues to gain a better understanding of battered women's cognitive states during counseling.
PRIME-MD Patient Health Questionnaire (PHQ-9) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Depression measure.
SPAN (Startle, Physiological arousal, Anger and Numbness) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Post-Traumatic Stress Disorder measure.
The SF-12 (v. 2) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Mental and Physical Health
The TWEAK | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Screening tool for alcohol abuse/dependency.
Drug Abuse Screening Tool (DAST) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Prescription and Street Drug Use.
The Intimate Partner Violence Strategies Index (IPV Strategies) | Baseline, 3-, 6-,12-, 18-, and 24-month postpartum
  Specific actions women take to cope with violence.
The Childhood Experiences of Violence Questionnaire Short Form (CEVQ-SF) | 6-month postpartum
  Childhood maltreatment
The Childhood Trauma Questionnaire (CTQ) | 6-month postpartum
  Childhood maltreatment.
A modified version of the Health and Social Service Utilization questionnaire | 6-,12-, 18-, and 24-month postpartum
  Assessment of service utilization.
Child health outcomes | Outcomes 1 and 2 are assessed at infant birth, 3 to 7 will be assessed at 6-, 12-, 18-, 24-month postpartum
  Data regarding the following child health outcomes are gathered by maternal interview: 1) birth weight; 2) length of gestation; 3) injuries; 4) emergency department visits (including those that are injury-related); 5) hospitalizations; 6) immunizations; and 7) developmental delay.
Child Protection Service records | 24-month postpartum
  Number of reports made, cases of confirmed child maltreatment, the type of maltreatment, the duration that cases were open, and whether children were placed in foster care or in custody of another family member.
The Public Health Nurses' Responses to Women Who Are Abused | Collected from nurses at baseline, 12 and 24 months
  Nurses' readiness to treat IPV. In the 20-item PHNR, nurses respond to one of two scenarios that resemble real-life experiences they would encounter in a postpartum home visit. The instrument measures nurses' thoughts, feeling and actions in response to identifying and responding to IPV. The PHNR has good internal consistency with an overall Cronbach alpha of 0.79.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet MacMillan, MD, Principal Investigator — McMaster University
Locations (1):
- 600 S. Commonwealth Ave., #800, Los Angeles, California, United States

REFERENCES:
- [Derived] Kalra N, Hooker L, Reisenhofer S, Di Tanna GL, Garcia-Moreno C. Training healthcare providers to respond to intimate partner violence against women. Cochrane Database Syst Rev. 2021 May 31;5(5):CD012423. doi: 10.1002/14651858.CD012423.pub2. PMID 34057734
- [Derived] Jack SM, Boyle M, McKee C, Ford-Gilboe M, Wathen CN, Scribano P, Davidov D, McNaughton D, O'Brien R, Johnston C, Gasbarro M, Tanaka M, Kimber M, Coben J, Olds DL, MacMillan HL. Effect of Addition of an Intimate Partner Violence Intervention to a Nurse Home Visitation Program on Maternal Quality of Life: A Randomized Clinical Trial. JAMA. 2019 Apr 23;321(16):1576-1585. doi: 10.1001/jama.2019.3211. PMID 31012933